CLINICAL TRIAL: NCT07381816
Title: GastroFlow: Investigation of the Gastrointestinal Blood Flow in Patients With Postprandial Hypotension
Acronym: Gastroflow
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: H-25007666; NNF23OC0082437 (Other Grant/Funding Number: Novo Nordisk Foundation)
Record Dates: First submitted 2025-09-03; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-09

CONDITIONS: Postprandial Hypotension; Healthy; Blood Flow
Keywords: Physiology; GIP; Blood flow; Postprandial hypotension; Splanchnic blood flow; Mesenteric blood flow
MeSH Terms: interventions — Magnetic Resonance Spectroscopy; Equipment and Supplies; Sodium Chloride; Glucose

STUDY DESIGN:
Intervention Model Description: Single blind, placebo controlled, randomized, crossover study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postprandial hypotension group (Experimental): MRI scans of PPH patients. 3 interventions
  Interventions: Other: MRI + GIPR antagonist (Tool); Other: MRI + hangrip; Other: Saline and oral glucose
- Healthy matched controls (Placebo Comparator): MRI scans of healthy controls. Crossover design three interventions.
  Interventions: Other: MRI + GIPR antagonist (Tool); Other: MRI + hangrip; Other: Saline and oral glucose

INTERVENTIONS:
Other: MRI + GIPR antagonist (Tool) — GIP(3-30)NH2 infusion, oral glucose during MRI scans
Other: MRI + hangrip — Hangrip exercises, oral glucose during MRI scans
Other: Saline and oral glucose — Saline infusion oral glucose during MRI scans

SUMMARY:
This project will describe the mechanisms of action and the relative contributions of GIP to changes in gastrointestinal blood flow induced by oral glucose and endogenous GIP with the use of a receptor antagonists GIP(3-30)NH2 in patients with postprandial hypotension.

DETAILED DESCRIPTION:
Each participant will attend three independent randomised experimental days in the MRI-scanner with intravenous infusion (hormone/placebo) and oral ingestion (glucose): An intravenous infusion of saline or GIP(3-30)NH2 starts at time point -20 minutes.The infusions are combined with an oral glucose tolerance test (75 gram of glucose dissolved in 250 ml water ingested orally) at time point 0 minutes on two of the experimental days (with and without GIP(3-30)NH2). Furthermore one day will be with handgrip exercise, without an infusion. Therefore the first two days are in randomized order.

MRI measurements are repeatedly performed and blood samples are drawn to be analysed for endocrine responses from the intestines and pancreas.

ELIGIBILITY:
For the PPH group

Inclusion Criteria:

* Postprandial hypotension
* Symptoms of postprandial hypotension

Exclusion Criteria:

* Treatment with drugs that cannot be paused for 12 hours
* Metallic implants that does not tolerate MRI
* Any other disease or dysfunction that may disturb blood flow to the gut
* Intake of more than 14 units of alcohol per week or abuse of drugs
* Blood vessels that are not feasible for measuring flow in the MRI scanner
* Low blood percent
* Decreased kidney function
* Decreased liver function
* Claustrophobia

For the healthy group

Inclusion Criteria:

* Matched by age, gender and BMI

Exclusion Criteria:

* Postprandial hypotension
* Metallic implants that does not tolerate MRI
* Intake of more than 14 units of alcohol per week or abuse of drugs
* Blood vessels that are not feasible for measuring flow in the MRI scanner
* Low blood percent
* Decreased kidney function
* Decreased liver function
* Claustrophobia
* Autonomic dysfunction or other disease that cause changes in blood pressure during or after a meal
* Intake of pharmaceutical products that influence the blood pressure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Blood flow | 145 minutes
  Redistribution of splanchnic blood flow in the vessel mesenteric superior artery. Measured with functional MRI in ml/min

SECONDARY OUTCOMES:
Blood flow | 145 minutes
  Blood flow in vena portae
Blood flow | 145 minutes
  Blood flow in trunks coeliacus

CONTACTS AND LOCATIONS:
Locations (1):
- Glostrup hospital, Glostrup Municipality, Denmark

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-15): https://cdn.clinicaltrials.gov/large-docs/16/NCT07381816/Prot_SAP_000.pdf